CLINICAL TRIAL: NCT05921747
Title: The Impact of Innovative Technology Strategies on Implementing Exercise Programs Using Fully Immersive Virtual Reality for Postpartum Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSAHS 2023/01
Record Dates: First submitted 2023-04-17; First posted 2023-06-27 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Post Partum Lumbopelvic Pain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: After selecting the desired sample size (tentative 17) the subjects will be randomly allocated to the both treatment groups
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants consented to participate will be assigned a unique number. The detailed list will be kept confidentially under the custody of the Principal Investigator. Unique numbered envelop will be provided to the participant. The participant will tell his number to the receptionist. The receptionist will send the participant to treatment room according to randomly allocation list. An outcome assessor will fill the form after treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional exercises as control group (Other): Traditional exercise as control group
  Postpartum women in this group will receive an 18-minute training session that will start with pelvic floor muscle training with 3 sets of 12 repetitions of 3 seconds of contraction and 3 seconds of relaxation in a lying position. The second part will be performed with 2 sets of 5-minute training modules with 1-minute rest between modules. A five-exercise circuit will be performed with one minute per exercise where the aim is to achieve the maximum number of repetitions possible, and then move on to the next exercise. For the exercises 2 dumbbells of 1 kilogram will be required. The exercises will include Kegel pelvic floor exercise, dead weight lifts, wide back rows, lunges with rotation, good morning (hip hinge), and lateral side bends. These traditional exercises were designed to build strength and improve pelvic floor function, lumbo-pelvic pain mirroring under the supervision of physiotherapist.
  Interventions: Other: Traditional exercise as control group
- VR Intervention Group Protocol (Experimental): Experimental: Participants in the intervention group will undergo a virtual reality (VR)-based exercise program using Meta Quest 2 head-mounted displays (Meta Platforms Inc., USA) and the Lumbar Pain Rehab software provided by DynamicsVR (Dynamics VR S.L., Cadiz, Spain). The virtual reality (VR) intervention will consist of eight structured sessions designed to address postpartum lumbo-pelvic pain through the immersive, interactive training.
  Each session incorporating pelvic floor muscle training using VR, consisting of three sets of 12 repetitions, with each contraction and relaxation phase lasting three seconds. In addition, patients engaged in two five-minute blocks of immersive VR activities with a two-minute rest interval, resulting in total session duration of 18 minutes.
  Interventions: Other: Traditional exercise as control group; Device: VR Intervention Group Protocol

INTERVENTIONS:
Other: Traditional exercise as control group — Standard Traditional exercise program:
  The traditional exercises will include Kegel pelvic floor exercise, dead weight lifts, wide back rows, lunges with rotation, good morning (hip hinge), and lateral side bends. .
  Pre and post measurement will be taken before and after the session.
Device: VR Intervention Group Protocol — Participants in the intervention group will undergo a virtual reality (VR)-based exercise program using Meta Quest 2 head-mounted displays (Meta Platforms Inc., USA) and the Lumbar Pain Rehab software provided by DynamicsVR (Dynamics VR S.L., Cadiz, Spain). The virtual reality (VR) intervention will consist of eight structured sessions designed to address postpartum lumbo-pelvic pain through the immersive, interactive training.
  Each session incorporating pelvic floor muscle training using VR, consisting of three sets of 12 repetitions, with each contraction and relaxation phase lasting three seconds. In addition, patients engaged in two five-minute blocks of immersive VR activities with a two-minute rest interval, resulting in total session duration of 18 minutes.
  A familiarization session will be conducted prior to the intervention to acclimate participants to the VR environment. This will include modified pelvic floor training (3 sets of 8 repetitions; 3 seconds of contraction.
  Other Names: VR Intervention Group Protocol as experimental group
  Arms: VR Intervention Group Protocol

SUMMARY:
The study aims to determine the effect of traditional exercise through using fully immersive virtual reality in postpartum female with lumbopelvic pain.

This study will be single-blind randomized clinical -trial and will be conducted at Shalamar Institute of health sciences in 1 year after the approval by institutional review board. Sixty female participants with a history of lumbopelvic pain will be recruited on the basis of inclusion and exclusion criteria. Data will be collected after taking written Informed Consent from each patient. The included participants will be randomized by gold fish randomization method and allocated to two groups (A & B) each with 30 participants.

DETAILED DESCRIPTION:
Lumbopelvic pain refers to self-reported pain in the lower back, sacroiliac joints, or a combination of these locations, among pregnant and postnatal women. Approximately 50% of pregnant women report lumbopelvic pain to some degree. Recent studies indicate the importance of hip extensors, pelvic floor muscle (PFM) and transverse abdominal muscle (TrAM) in the development of lumbopelvic pain.Moreover, pelvic instability, asymmetry and insufficient compression of the sacroiliac joints contribute to continuous lumbopelvic pain after delivery. In Europe every tenth women shortly postpartum and every sixth has reported similar symptoms 6 weeks later. Age, PGP during pregnancy and abdominal midline doming were associated with experiencing PGP shortly postpartum.

Studies have demonstrated the importance of choosing an optimal treatment strategy in clinical practice, and 5 subgroups of self-rated pain locations have been identified in the pelvic area. The study focused on pelvic girdle pain (PGP), or PGP in combination with lumbar pain, since these groups have been shown to have the highest impact on activity levels and health-related quality of life.

Traditional exercises that include dynamically controlling the lumbar segments and pelvic joints have been shown to result in functional improvement in patients with lumbopelvic pain. The term "core stability" is commonly used to refer to the ability of these "core" muscles to stabilize the lumbar spine and pelvic girdle during static postures and dynamic movements. A host of theories and "stabilization exercise" programs have been developed to train these muscles as a means of treating and/or preventing lower back pain (LBP). However, there is still much inconsistency and debate both in the clinical and research communities with regards to what constitutes "core stability" and a "stabilization exercise". Chronic pain is a global healthcare burden with as much as of 11% of the US population suffering from pain lasting six months or longer, and upwards of 20% in Europe. Chronic pain can lead to depression, anxiety, sleep disturbances, and impairment in cognitive tasks.

Established research supports VR(virtual relaity) as a treatment strategy for burn pain, acute pain, and experimentally induced pain. Two primary approaches afford analgesic benefits of VR: distraction therapy and immersive-ness. Distraction therapy temporarily takes attention away from pain while patients are engaged in the VR experience. In immersive VR, the user can interact with an artificial environment to treat chronic pain. In immersive VR, the user can interact with an artificial environment to treat chronic pain. One form of immersive VR is virtual embodiment. Virtual embodiment refers to the sense of owning a virtual body, from a first-person perspective, feeling the agent of the sensory feedback related to the actions of the virtual body. Through activation of somatosensory and premotor circuitry associated with the body parts that are embodied, the use of virtual embodiment as an immersive VR technique has been shown to influence pain-free range of motion in patients with unilateral chronic shoulder pain.

A case series was conducted in 2020, in which they describe two case studies that use embodiment in virtual reality as a treatment for chronic low back pain. The purpose of this case series was to determine the feasibility of a novel virtual reality-based digital therapeutic for the treatment of chronic pain. Two patients with chronic low back pain received seven sessions, two sessions per week, of a novel digital therapeutic that combines virtual embodiment with graded motor imagery to deliver functional rehabilitation exercises using an off-the-shelf virtual reality system. Pain catastrophizing scale was assessed before the first session and after the seventh session to determine the extent to which virtual embodiment training can improve psychological symptoms of chronic low back pain. In both patients, pain intensity was improved after individual sessions of virtual embodiment training. They concluded that embodiment in virtual reality improves symptoms of persistent chronic low back pain.

A study (RCT) was conducted in 2022 and their study have measured the Effects of a motor control exercise program on lumbopelvic pain recurrences and intensity in pregnant women with a history of lumbopelvic pain. Forty pregnant women with a history of lower back pelvic pain (LBPP) were recruited and randomly allocated to a control (20 participants) or intervention (20 participants) group. The control group have received standard prenatal care, including basic information on what to do when suffering from LBPP. The intervention group have participated in three 40-min exercise sessions per week from < 20 weeks until 34-36 weeks of gestation: one supervised group session via the Zoom platform (once a month) and two unsupervised sessions at home. A motor control exercise program was developed to target strengthening of the lumbo-pelvic-hip core muscles and to improve spinal and pelvic stabilization. Participants of this group have also received standard prenatal care. They concluded that motor control exercise program have allowed pregnant women to progress at their own pace through different levels of exercises. In addition, the use of technology in the follow-up of the women will make the approach flexible and adapted to their daily routines.

The purpose of the study is to reduce the potential abuse, dependency of painkillers and manual therapy intervention for treating chronic lumbopelvic pain. In order to promote an advance and noninvasive method for treating lumbopelvic pain in postpartum female this study will help to design better rehabilitative program including core stability exercise using the analgesic and distracting effects of Immersive Virtual reality. This study will help physiotherapist as well as other health care professionals to treat other factors contributing to lumbopelvic pain other than weak muscles and posture alignment in postpartum female through virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women with acute and chronic lumbopelvic pain.
* Primary parous & multiparous women.

Exclusion Criteria:

* Postpartum women with nausea, dizziness and blurred vision, high risk pregnancies.
* Structural disorder of spinal alignment (Scoliosis, kyphosis, lordosis)
* Traumatic/ Inflammatory / Infectious Conditions
* Diagnosed stress / depression
* History of spinal, pelvic, or femur surgery or previous fracture, neoplasm
* Any Previous history of backache

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Post partum Female
Enrollment: 34 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
Effect on lumbopelvic pain | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  During pregnancy, women go through several hormonal and biomechanical changes as well as neuromuscular adaptations which could explain the development of lumbopelvic pain. Pregnancy-related hormonal changes, characterized by an increase in relaxin, estrogen and progesterone levels, are potentially linked to hyperlaxity of ligament and joint instability, thus contributing to lumbopelvic pain. In addition, biomechanical changes induced by the growing fetus, can modify posture, load sharing and mechanical stress in the lumbar and pelvic structures. Finally, neuromuscular adaptations during pregnancy include an increase in the activation of lumbopelvic muscles and a decrease in endurance of the pelvic floor muscles. Short Form McGill Pain Questionnaire(SF-MPQ) will be used to determine the intensity of pain.
  The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Effect on disability due to lumbopelvic pain | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  Due to physiological changes the pregnant female experience lumber pain. to determine lumber pain Oswestry Disability Index (ODI) will be used.
  ODI scale will include following levels for assessment 0 - 4 No disability 5 - 14 Mild disability 15 - 24 Moderate disability 25 - 34 Severe disability 35 - 50 Completely disabled
Effect on disability due to pelvic pain | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  Pelvic Floor Disability Index ( PFDI) will be used to assesses the distress of pelvic organ prolapse (POP), anorectal and urinary symptoms in three subscales, respectively, Pelvic Organ Prolapse Distress Inventory (POPDI-6), Colorectal-Anal Distress Inventory (CRADI-8) and Urinary Distress Inventory (UDI-6) .The PFDI-20 has 20 items and 3 scales of your symptoms. All items use the following format with a response scale from 0 to 4. Scale Scores
Effect on functioning | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  Patient Specific Functional Scale(PSFS) will be used. This scale will nominate 3 to 5 activities that they are unable to do or having difficulty doing because of their injury or problem. These activities are rated on an 11-point scale, where 0 is unable to perform the activity and 10 is able to perform the activity at preinjury level.
Level of Depression, anxiety & stress | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  DASS (Depression anxiety stress scale)questionnaire will be used for assessment. The total score represents overall distress (0 to 30), with higher scores indicating more severe distress or a greater number of symptoms. Two subscales are presented: Anxiety-Stress: Items 1, 4, 6, 7, 8, 9 (raw score range = 0 to 18) Depression: Items 2, 3, 5, 10 (raw score range = 0 to 12)
To access intensity of Pain | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  Visual analog scale (VAS) will be used to determine the intensity of pain. The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
condition-specific measure for women with pelvic girdle pain | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  Pelvic Girdle Questionnaire (PGQ) will be used .To calculate the total PGQ score, all scores are summarized and divided by the total possible score of 75 (maximum possible scores of 60 for activity and 15 for symptoms), subsequently recalculated to a percentage, resulting in percentage scores ranging from 0 (no disability) to 100 (severe disability).

SECONDARY OUTCOMES:
Level of Urinary incontinence | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  Urinary Distress Index will be used to access distress caused by urinary incontinence.UDI-6 scores more than 33.33 indicate higher distress caused by urinary incontinence symptoms.
To access fear of movement | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  Tampa scale of kinesiophobia (TSK). TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia
Psychological assessment (Rumination, Magnification &Helplessness) | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  Pain Catastrophizing Scale will be used for measurement. Patients are asked to rate the degree to which they have any of the thoughts described in the questionnaire using a 5-point Likert scale ranging from 0 (never) to 4 (always). The total score is the sum of the scores for the individual items, and ranges from 0 to 52.

OTHER OUTCOMES:
Presence of Vestibular basilar artery insufficiency (VBI) | Pre Treatment one time (Day 0)
  VBI test will be performed for assessment. Test is considered positive if there is dropping of the arms, loss of balance, or pronation of the hands; a positive result indicates decreased blood supply to the brain.
  If it turns out positive then patient wont be included in the research due to use of Virtual reality.
Presence of Simulator Sickness | Baseline (Day 0) , Follow up 1 (Day 30) after 8 sessions of treatment and follow up 2nd (day 60).
  Simulator Sickness Questionnaire (SSQ) will be used for assessment .The overall support score (SSQN) is calculated by taking an average of the individual scores across the 27 items. A high score on the SSQ indicates more optimism about life than a low score. Respondents with low SSQ scores have a higher prevalence of negative life events and illness.

CONTACTS AND LOCATIONS:
Overall Officials: Javeria Dr Aslam, Ph.D, Principal Investigator — Shalamar Institute of Health Sciences; Carlos R. Morales, Ph.D, Study Director — Universided Europea Madrid, Spain; RAQUEL DIAZ-MECO, Ph.D, Study Director — Universided Europea Madrid, Spain; Alba P. Alemany, Ph.D, Principal Investigator — Department of Radiology & Physical Medicine, Complutense University of Madrid, Spain
Locations (1):
- Shalamar School of Allied Health Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vesentini G, Prior J, Ferreira PH, Hodges PW, Rudge M, Ferreira ML. Pelvic floor muscle training for women with lumbopelvic pain: A systematic review and meta-analysis. Eur J Pain. 2020 Nov;24(10):1865-1879. doi: 10.1002/ejp.1636. Epub 2020 Sep 6. PMID 32735717
- [Background] Daneau C, Abboud J, Marchand AA, Houle M, Pasquier M, Ruchat SM, Descarreaux M. Mechanisms Underlying Lumbopelvic Pain During Pregnancy: A Proposed Model. Front Pain Res (Lausanne). 2021 Dec 2;2:773988. doi: 10.3389/fpain.2021.773988. eCollection 2021. PMID 35295430
- [Background] Catena RD, Wolcott WC. Self-selection of gestational lumbopelvic posture and bipedal evolution. Gait Posture. 2021 Sep;89:7-13. doi: 10.1016/j.gaitpost.2021.06.022. Epub 2021 Jun 26. PMID 34217002
- [Background] Starzec-Proserpio M, Wegrzynowska M, Sys D, Kajdy A, Rongies W, Baranowska B. Prevalence and factors associated with postpartum pelvic girdle pain among women in Poland: a prospective, observational study. BMC Musculoskelet Disord. 2022 Oct 20;23(1):928. doi: 10.1186/s12891-022-05864-y. PMID 36266709
- [Background] Trujillo MS, Alvarez AF, Nguyen L, Petros J. Embodiment in Virtual Reality for the Treatment of Chronic Low Back Pain: A Case Series. J Pain Res. 2020 Nov 25;13:3131-3137. doi: 10.2147/JPR.S275312. eCollection 2020. PMID 33269003
- [Background] Luo Y, He L, Li Y, Xie J, Gong S, Zhang Q, Yin E, Gu M, Yi C. Sacral osteotomy combined with triangular osteosynthesis in the treatment of malunion and nonunion of vertically displaced pelvic fractures. J Orthop Surg Res. 2022 Sep 5;17(1):409. doi: 10.1186/s13018-022-03296-x. PMID 36064584
- [Background] Beales D, Lutz A, Thompson J, Wand BM, O'Sullivan P. Disturbed body perception, reduced sleep, and kinesiophobia in subjects with pregnancy-related persistent lumbopelvic pain and moderate levels of disability: An exploratory study. Man Ther. 2016 Feb;21:69-75. doi: 10.1016/j.math.2015.04.016. Epub 2015 May 1. PMID 25997987
- [Result] Saleh MSM, Botla AMM, Elbehary NAM. Effect of core stability exercises on postpartum lumbopelvic pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(2):205-213. doi: 10.3233/BMR-181259. PMID 30282349
- [Result] Ehsani F, Sahebi N, Shanbehzadeh S, Arab AM, ShahAli S. Stabilization exercise affects function of transverse abdominis and pelvic floor muscles in women with postpartum lumbo-pelvic pain: a double-blinded randomized clinical trial study. Int Urogynecol J. 2020 Jan;31(1):197-204. doi: 10.1007/s00192-019-03877-1. Epub 2019 Apr 23. PMID 31016337
- [Result] Sonmezer E, Ozkoslu MA, Yosmaoglu HB. The effects of clinical pilates exercises on functional disability, pain, quality of life and lumbopelvic stabilization in pregnant women with low back pain: A randomized controlled study. J Back Musculoskelet Rehabil. 2021;34(1):69-76. doi: 10.3233/BMR-191810. PMID 32986655
- [Result] Matamala-Gomez M, Slater M, Sanchez-Vives MV. Impact of virtual embodiment and exercises on functional ability and range of motion in orthopedic rehabilitation. Sci Rep. 2022 Mar 23;12(1):5046. doi: 10.1038/s41598-022-08917-3. PMID 35322080
- [Result] Daneau C, Marchand AA, Bussieres A, O'Shaughnessy J, Ruchat SM, Descarreaux M. Effects of a motor control exercise program on lumbopelvic pain recurrences and intensity in pregnant women with a history of lumbopelvic pain: a study protocol for a randomized controlled feasibility trial. Pilot Feasibility Stud. 2022 Mar 21;8(1):65. doi: 10.1186/s40814-022-01024-0. PMID 35313988
- [Result] Kale, A.A. and Pathan, N.M., 2019. Effect of Core Stabilisation Exercises in Postnatal Women with Lumbo-Pelvic Instability. Indian Journal of Physiotherapy and Occupational Therapy, 13(2), p.19.